CLINICAL TRIAL: NCT05289193
Title: CD8+ Cell Imaging During Neoadjuvant ImmunoTherapy (The C-IT Neo Trial)
Brief Title: CD8+ T Cell Imaging During Pre-surgery Immunotherapy in People With Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-456
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Melanoma; Melanoma Stage III
Keywords: CD8+ Cell Imaging; C-IT Neo Trial; stage III melanoma; 89Zr-Df-Crefmirlimab; Memorial Sloan Kettering Cancer Center; 21-456
MeSH Terms: conditions — Melanoma | interventions — Positron-Emission Tomography; Nivolumab; Ipilimumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with Stage III Melanoma (Experimental): All participants will have cytologically or histologically confirmed stage IIIB, IIIC, IIID melanoma that can be surgically removed.
  Interventions: Diagnostic Test: PET Scan; Drug: Nivolumab; Drug: Ipilimumab; Procedure: Surgical Resection of Melanoma

INTERVENTIONS:
Diagnostic Test: PET Scan — Patients will have a baseline CD8 PET scan prior to one dose of neoadjuvant nivolumab
  1mg/kg + ipilimumab 3mg/kg. After 4 weeks, patients will have a repeat CD8 PET scan and then undergo surgical resection of their stage III melanoma.
  Other Names: 89Zr-Df-Crefmirlimab
Drug: Nivolumab — Patients will have a baseline CD8 PET scan prior to receiving one dose of neoadjuvant nivolumab
  1mg/kg + ipilimumab 3mg/kg.
Drug: Ipilimumab — Patients will have a baseline CD8 PET scan prior to receiving one dose of neoadjuvant nivolumab
  1mg/kg + ipilimumab 3mg/kg.
Procedure: Surgical Resection of Melanoma — Patients will have a baseline CD8 PET scan prior to one dose of neoadjuvant nivolumab
  1mg/kg + ipilimumab 3mg/kg. After 4 weeks, patients will have a repeat CD8 PET scan and then undergo surgical resection of their stage III melanoma.

SUMMARY:
Combination treatment with nivolumab and ipilimumab before surgery may help people with melanoma because the drugs are designed to help the immune system target and destroy cancer cells (immunotherapy), which may shrink the cancer and prevent recurrence after surgery. Treatment given before surgery is called neoadjuvant therapy. The purpose of this study is to find out whether neoadjuvant therapy with nivolumab and ipilimumab can kill melanoma tumors before surgery and prevent disease from coming back after surgery. This study also explores a new, experimental PET scan that images the immune system to see if it is related to treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patient is capable of understanding and complying with the protocol requirements and has signed the Informed Consent document.
* Adults at least 18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Cytologically or histologically confirmed stage IIIB, IIIC, IIID, or IV melanoma that can be surgically removed.

Notes:

* In-transit melanoma is acceptable.
* Patients can enroll regardless of their BRAF mutational status

  * 1cm of tumor needs to be visible on standard imaging (i.e. FDG PET or CT scan)
  * Screening laboratory values must meet the following criteria:
* WBC ≥ 2.0x109/L
* Neutrophils ≥ 1.5x109/L
* Platelets ≥ 100 x109/L
* Hemoglobin ≥ 5.5 mmol/L
* Creatinine ≤ 1.5x ULN
* AST ≤ 1.5 x ULN and ALT ≤ 1.5 x ULN
* Bilirubin ≤1.5 X ULN

  * Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception. WOCBP should use an adequate method to avoid pregnancy for 23 weeks (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of study treatment (ipilimumab/nivolumab)
  * Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of ipilimumab + nivolumab
  * Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year. Men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of study treatment (ipilimumab/nivolumab)

Note: Women who are not of childbearing potential (i.e., who are postmenopausal), or surgically sterile as well as azoospermic men do not require contraception

Exclusion Criteria:

* Subjects with any active autoimmune disease (current symptoms or requirement for immunosuppression at the time of study start).
* Positive active hepatitis B viral infection (+viral load by PCR)
* Prior immunotherapy targeting CTLA-4 and/or PD-1/PD-L1 for any disease.
* Potentially unresectable melanoma.
* History of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* History of severe hypersensitivity reaction to any monoclonal antibody
* Underlying medical conditions that, in the Investigator's opinion, will make the administration of treatment hazardous or obscure the interpretation of toxicity
* Patients who have undergone splenectomy or have other splenic disorders. The normal spleen usually has CD8+ cell activity and serves as a positive control to enable proper imaging technique.
* Use of other investigational drugs before study drug administration 30 days and 5 half-times before study inclusion
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2026-03-11 (Estimated); Study Completion 2026-03-11 (Estimated)

PRIMARY OUTCOMES:
Major pathologic responses/MPR | up to 2 years
  Participants' disease will be assessed for MPR as per previously established criteria for neoadjuvant trials (near complete response ≤10% viable; complete response 0% viable). Pathologic response (≤50% viable) will also be estimated.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Postow, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org